CLINICAL TRIAL: NCT04798404
Title: Integrating a Prevention Care Path Into Daily Life of Elders With Mobility Disability Risk: Introducing a Predictive Model to a Functional Exercise Response
Brief Title: Integrated Care Analysis Response to Exercise in Community-dwelling Elders
Acronym: ICARE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1091
Record Dates: First submitted 2021-02-23; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Physical Activity; Gerontology
Keywords: elders; mobility; prevention; predictive model; resistance training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exercise Intervention in 20 collective sessions: 104 elders recruited among the community (mean age: 82.1 ± 5.7, 72 women and 32 men), diagnosed in initial consultation with mobility disability risk (sedentary or/and pre-frail/frail or/and sarcopenia at least probable) who participated in 20 collective sessions twice a week and two hours per week, and have been seen for reassessment in final consultation.
  Interventions: Other: Multimodal exercise intervention

INTERVENTIONS:
Other: Multimodal exercise intervention — The intervention conducted was a progressive multicomponent training protocol. The training consisted on 2 collective sessions of 1h per week, during 10 weeks. Sessions involved functional exercises, muscular reinforcement performed at body-weight or with small materials (elastic bands or dumbbells), balance, and adapted sport and physical activities. Progression was based on an increase in workload (or in muscle strains). The workload was considered as the interaction of intensity and volume of exercise (set x repetitions). Intensity was based on effort tolerance, modulate by contraction regimen, velocity and load (elastic bands stiffness). Participants were encouraged to reproduce exercises at home when they were performed easily in supervised collective sessions.

SUMMARY:
One of the main challenges of ageing is to prevent the onset of mobility disability and its co-morbidities. Screening the risk of mobility disability in community-dwelling elders is therefore very important and at the uppermost for the care of sarcopenia and frailty. A multicomponent intervention, integrating multidisciplinary actions and combining physical exercise and nutrition, is recognized as an effective therapy for the care of mobility disability risk factors. The diagnosis of either pre-frail/frailty and/or sarcopenia at least probable is sufficient to trigger a sustained intervention as it can prevent the onset of mobility disability. Therefore, it is difficult to identify the best responder for this type of care path. As a result, studies have been interested in exploring the predictive factors related to the functional response to exercise within lifestyle interventions. It has been shown that SPPB provides useful information when associated with demographic or physical activity factors. Those predictions are reliable to an ageing population with a SPPB ≤9 but it is still unknown if these reports are reproducible to older adults with high baseline physical function. Therefore, we hypothesized that a more inclusive SPPB score at baseline could also be related to other factors to predict the functional response to exercise. We assumed that strength, age, sex or body mass index could be interesting to elicit better predictions. It is an important issue for the development of targeted-interventions and specific care orientations.

The training has to be established through an accurate schedule to optimize the response to exercise. However, it is difficult to make consensus on the best method to apply, especially for elders with mobility disability risk. Hence, the present study also focus on a specific training method planned toward different exercises modes. We aimed to propose a training with cost-effective material and the absence of machines to transpose it into daily life participants. We expected to observe benefits on physical performance after this exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 70 years old
* Diagnosed with mobility disability risk during the initial assessment (sedentary or/and pre-frail/frail or/and sarcopenia at least probable)
* Have completed the 20 collective sessions
* Have been reassessed after 3 months of intervention

Exclusion Criteria:

* Baseline SPPB < 5
* Erroneous clinical data

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling elders diagnosed with risk mobility disability risk and who participated in 20 collective sessions of resistance training.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (score /12) | Change in the SPPB score at 3 months of intervention
  The use of SPPB is widely recognized for its ability to accurately assess the risk of mobility disability in elderly. It is based on the result of three assessments; static balance test, the ability to perform five chair lifts as quickly as possible and a walking speed test measured over four or six meters. SPPB give a score for 0 to 12 with an increased risk of mobility disability for a score less or equal to 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France